CLINICAL TRIAL: NCT01191632
Title: Randomised Controlled Phase I/II Trail to Evaluate the Effect of Neoadjuvant Radiation on Tumor Infiltrating T-cells by Low Dose Radiation Therapy in Resectable Colorectal Liver Metastases Patients
Brief Title: Effect of Neoadjuvant Radiation on Tumor Infiltrating T-cells by Low Dose Radiation in Colorectal Liver Metastases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Juergen Weitz, Department of surgery, university of Heidelberg
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S081/2008
Record Dates: First submitted 2010-08-20; First posted 2010-08-31 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Colorectal Liver Metastases
Keywords: T cell; surgery; radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Radiation 0,5Gy (Active Comparator): Radiation: one time Radiation with an intensity of 0.5 Gy Group A
  Beginning on a weekday 48 hours before surgery
  Interventions: Radiation: one time radiation
- No radiation (Active Comparator): Control group with 0Gy radiation
  Interventions: Radiation: No Radiation
- Radiation 2Gy (Active Comparator): Radiation: one time Radiation with an intensity of
  2.0 Gy Group B
  Beginning on a weekday 48 hours before surgery
  Interventions: Radiation: one time radiation
- Radiation 5Gy (Active Comparator): Radiation: one time Radiation with an intensity of
  5 Gy Group C Beginning on a weekday 48 hours before surgery
  Interventions: Radiation: one time radiation

INTERVENTIONS:
Radiation: one time radiation — Radiation: one time Radiation with an intensity of
  0.5 Gy Group A 2.0 Gy Group B 5 Gy Group C Beginning on a weekday 48 hours before surgery
  Arms: Radiation 0,5Gy; Radiation 2Gy; Radiation 5Gy
Radiation: No Radiation — Control group with 0Gy
  Arms: No radiation

SUMMARY:
The efficiency of T cell based immunotherapies is affected by the insufficient migration and activity of tumor specific effector T cells in the tumor. Aim of this phase I/II clinical trial is to evaluate whether a neoadjuvant, low dose radiotherapy can improve T cell connected anti tumor immune response in colorectal liver metastases.

The primary endpoint is the number of tumor infiltrating T cells. Furthermore the T cell activity in situ, the number of regulatory T cells and the frequency of tumor reactive T cells in the blood and bone marrow will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)
* Age ≥ 50 years
* Radiological urgently suspected colorectal liver metastasis

Exclusion Criteria:

* second malignancy
* Pregnancy and lactation
* no prior liver radiation
* liver metastasis must be resectable

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Purpose of the study is the determination of an active local external beam radiotherapy dose leading to a maximal number of tumor infiltrating T-cells. The total T-cell activity serves as primary surrogate parameters for anti- tumor activity | 2 years

SECONDARY OUTCOMES:
To determine local control and recurrence patterns of colorectal liver metastases in a CT | 2 years
To determine the progression-free survival in patients treated with low dose photon beam radiation therapy | 2 years
• To determine the surgical morbidity in patients undergoing liver resection who received this protocol treatment | 2 years
• To determine 30-day post-operative mortality after liver resection in patients who received this protocol treatment | 2 years
• To determine the T-cell activity in the resected liver tissue | 2 years
• To determine quality of life according to the EORTC QoL questionnaire after 6 months. | 6 months
To determine the number of regulatory T-cells in the resected liver tissue | 2 years
To determine the frequencies of tumor-reactive T-cells in the blood and bone marrow of the patients | 2 years
To determine quality of life according to the EORTC QoL questionnaire after 12 months. | 1 year
To determine the number of patients with adverse events as a measure of safety and tolerability according to CTCAE, Version 4.0 criteria | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Reissfelder C, Timke C, Schmitz-Winnenthal H, Rahbari NN, Koch M, Klug F, Roeder F, Edler L, Debus J, Buchler MW, Beckhove P, Huber PE, Weitz J. A randomized controlled trial to investigate the influence of low dose radiotherapy on immune stimulatory effects in liver metastases of colorectal cancer. BMC Cancer. 2011 Sep 30;11:419. doi: 10.1186/1471-2407-11-419. PMID 21961577